CLINICAL TRIAL: NCT05709249
Title: Efficacy of Xian-Lian-Jie-Du Optimization Decoction As an Adjuvant Treatment for Prevention of Recurrence of Stage IIIB/IIIC Colon Cancer：a Study Protocol for a Randomized Controlled Trial
Brief Title: Xian-Lian-Jie-Du Optimization Decoction As an Adjuvant Treatment for Prevention of Recurrence of Colon Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Collaborators: Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022NL-203-02
Record Dates: First submitted 2023-01-17; First posted 2023-02-02 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Colon Cancer
Keywords: colon cancer; Traditional Chinese medicine
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): Subjects in the intervention group will be treated with XLJDOD compound granule.
  Interventions: Drug: XLJDOD compound granule
- control group (Placebo Comparator): Subjects in the control group will be treated with placebo (XLJDOD mimetic agent).
  Interventions: Drug: placebo (XLJDOD mimetic agent)

INTERVENTIONS:
Drug: XLJDOD compound granule — Treatment will begin within 3 months after standard adjuvant chemotherapy and compliance will be continuously monitored. XLJDOD will be taken twice a day, infused with warm water, 1 hour after lunch and dinner. One course of treatment will take 28 days in 1 month, and 2- to 3-day rest. Treatment will continue for 6 courses.
  Arms: intervention group
Drug: placebo (XLJDOD mimetic agent) — The course of placebo in control group will be in accordance with that of XLJDOD in intervention group.
  Arms: control group

SUMMARY:
This study is designed as a multi-center, randomized, double-blind, placebo-controlled trial. Subjects in the intervention group will be treated with XLJDOD compound granule. Subjects in the control group will be treated with placebo (XLJDOD mimetic agent).

DETAILED DESCRIPTION:
Subjects in the intervention group will be treated with XLJDOD compound granule. Treatment will begin within 3 months after standard adjuvant chemotherapy and compliance will be continuously monitored. XLJDOD will be taken twice a day, infused with warm water, 1 hour after lunch and dinner. One course of treatment will take 28 days in 1 month, and 2- to 3-day rest. Treatment will continue for 6 courses. Subjects in the control group will be treated with placebo (XLJDOD mimetic agent). The course of placebo in control group will be in accordance with that of XLJDOD in intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Colon carcinoma confirmed by pathology.*

   *Preoperative endoscopy showed that the distal end of the tumor was ≥12cm from the anal margin. If the patient did not undergo endoscopic examination before surgery, the distance of the tumor from the anal margin was ≥12cm according to the results of intraoperative examination or preoperative imaging examination.
2. Completion of surgical resection of tumors with negative margins (R0 resection) and at least 3 months of adjuvant chemotherapy based on 5-fluorouracil (5-FU). *

   *4 cycles of CAPOX (capecitabine and oxaliplatin), 6 cycles of FOLFOX (fluorouracil, leucovorin, and oxaliplatin) or 4 cycles of single agent-5-FU, etc.
3. Within 3 months after the completion of adjuvant chemotherapy.
4. Patients with Stage IIIB or IIIC disease.*

   *IIIB: T3-T4aN1/N1cM0, T2-T3N2aM0 and T1-T2N2bM0, IIIC: T4aN2aM0, T3-T4aN2bM0 and T4bN1-N2M0, as defined by the American Joint Committee on Cancer (AJCC) 8th edition).
5. Aged 20-80 years, men or women.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. With no radiographic evidence of tumor recurrence.
8. Sign the informed consent form.

Exclusion Criteria:

1. Presence of other malignancies in the past 5 years except curatively treated basal cell carcinoma or cervical carcinoma in situ.
2. Besides adjuvant chemotherapy, other adjuvant therapy such as radiotherapy, targeted therapy and immunotherapy has been used to treat colon cancer.
3. Antitumor Chinese patent medicine and decoction have been used for more than 3 months after surgery or within 1 month before enrollment.
4. Patients with severe comorbidities such as cardiovascular, cerebrovascular, renal, hepatic, hematopoietic system and other severe primary diseases.
5. Allergic to the ingredients of XLJDOD.
6. Any condition that is unstable or can jeopardize the safety of the patients and their compliance to the study, including pregnancy, plan to be pregnant, lactation and psychiatric disorders (schizophrenia, depression, and obsessive-compulsive disorder, etc.).
7. Suspected or confirmed history of alcohol and drug abuse.
8. Patients with other conditions considered by the investigator should not participate in the study.
9. Patients who have recently participated in or are currently participating in other clinical trials of drugs.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Two-year disease-free survival (DFS) | Assess once 24 months after randomization
  2-year DFS is defined as the percentage of patients alive without disease recurrence at 2 years measured from the randomization date.

SECONDARY OUTCOMES:
Three-year disease-free survival (DFS) | Assess once 36 months after randomization
  3-year DFS is defined as the percentage of patients alive without disease recurrence at 3 years measured from the randomization date.
One, two, three-year relapse rate (RR) | Assess at month 12, 24, 36 after randomization
  RR is defined as the fraction of followed patients who have disease recurrence. All disease recurrences and deaths from colon cancer are events. Second primary same cancers and other primary cancers will be ignored.
Three-year survival rate | Assess once 36 months after randomization
  3-year survival rate is defined as the percentage of patients alive at 3 years measured from the randomization date.
Overall survival (OS) | Observation to the end of the study，assessed up to 24 months
  OS is measured from the date of enrollment to the date of death, irrespective of cause.
Changes in total score on the EORTCQLQ-C30 Scale | Measurement will be performed at baseline and month 6, 12 ,18 ,24, 36.
  The changes of The European O-rganization for Reasearch and Treatment of Cancer score will be compared in the two groups prior to and following XLJDOD compound granule administration. It is a universal scale for all patients with malignant tumors with a total score of 126, ranging from 30 (least severe) to 126 (most severe).
Changes in total score on the MD Anderson Symptom Inventory for Traditional Chinese Medicine (MDASI-TCM) | Compared with the baseline period, the changes in MDASI-TCM score at month 6, 12 ,18 ,24, 36 will be measured.
  The scale is divided into two parts. The first part mainly assesses the severity of 20 common clinical symptoms and TCM-related symptoms of patients with cancer in the past 24 hours. The second part is the evaluation scale of the interference of the above symptoms with daily functioning. It has a total of 26 items, each with a score of 0-10, leading to a total score of 0-260.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Geng X, Wang Z, Feng L, Gu Y, Wang R, Yao Q, Xu Y, Wu J, Jiang Z, Chen K, Hu W, Tang D, Huo J, Li L, Bu Q, Zhao S, Zhang B, Cheng H. Efficacy and safety of Xian-Lian-Jie-Du optimization decoction as an adjuvant treatment for prevention of recurrence in patients with stage IIIB/IIIC colon cancer: study protocol for a multicentre, randomized controlled trial. BMC Complement Med Ther. 2023 Jul 17;23(1):239. doi: 10.1186/s12906-023-04052-2. PMID 37461034